CLINICAL TRIAL: NCT02282306
Title: Pilot Evaluation of the "Tailored Telephone Intervention Delivered by Peers to Prevent Recurring Opioid-Overdoses"
Brief Title: Phone Interview to Prevent Recurring Opioid Overdoses
Acronym: TTIP-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Theresa Winhusen, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-2591
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Overdose; Opioid-related Disorders; Drug Addiction; Drug Abuse; Substance Abuse; Opioid Use, Unspecified; Opioid Dependence; Drug Overdose
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TTIP-PRO (Other): Patients who have experienced an OOD in the past 8 months will be eligible to receive TTIP-PRO. A letter about the study will be sent to those patients. Interested patients will call the UC Health staff working on this study. The intervention entails administering the Personal Opioid-Overdose Risk Survey and the Opioid Overdose and Treatment Awareness Survey to the patient. The TTIP-PRO computer program uses the information to generate the "Personal Feedback Report", which is used by the Peer Interventionist to provide the intervention. The TTIP-PRO computer program also creates the "Personal Risk Factors Report" which is mailed to the participant with some other helpful information.
  Interventions: Behavioral: TTIP-PRO

INTERVENTIONS:
Behavioral: TTIP-PRO — The peer-delivered TTIP-PRO intervention is designed to: 1). increase the patient's knowledge of risk factors for OOD, with a particular emphasis on the patient's personal risk factors. This aim is one of harm reduction and is intended to help patients who continue to abuse opioids to use in a safer manner and 2).For patients who are open to considering treatment, to encourage the patient to get treatment for his/her opioid use disorder. This goal is based on research findings that effective treatment reduces the risk of OOD.

SUMMARY:
There has been a dramatic rise in opioid overdose (OOD) deaths in recent years. Attempts to ameliorate the problem have largely focused on increasing the accessibility of naloxone, an opioid antagonist that is effective in OOD reversal. Individuals who have experienced a non-fatal OOD are at risk for additional overdoses and yet there are no interventions that specifically target this high-risk population. To address this gap, the investigators have developed the "Tailored Telephone Intervention delivered by Peers to Prevent Recurring Opioid Overdoses" (TTIP-PRO). The overall goal of the present study is to conduct a pilot evaluation of the TTIP-PRO. The research literature suggests the need for an intervention targeting patients experiencing a non-fatal OOD.

DETAILED DESCRIPTION:
This is a single-group, unblinded pilot study of the TTIP-PRO, which will be completed with approximately 30 participants. Potential participants will be identified by querying the University of Cincinnati Medical Center (UCMC) Emergency Department (ED) Electronic Health Record (EHR) for patients treated for an OOD (e.g., opioid poisoning). Patients who have experienced an OOD in the past 8 months will be eligible to receive the TTIP-PRO. A letter about the study will be sent to those patients. Interested patients will call the UC Health staff working on this study. A UC Health staff member will inform potential participants about the study, confirm eligibility, collect enrollment measures, and schedule a time for the TTIP-PRO to be completed with the Peer Interventionist. The participant will be instructed to contact the Peer Interventionist at the scheduled time. After the peer-delivered TTIP-PRO intervention has been completed, a UC Health employee will contact the participant to administer the follow-up measures. The UC Health employee will then send a mailing to the participant that will include a copy of the participant's "Personal Risks for Overdose" report, general information about overdose prevention, and information about treatment for opioid use disorder (see section 2.6 for additional information). The mailing will also include a gift card (which is a standard part of the TTIP-PRO) and an additional gift card to compensate the participant for his/her time as a study participant.

ELIGIBILITY:
Inclusion Criteria for participants (receiving the TTIP-PRO intervention):

* have been treated for an OOD by the UCMC ED within the prior 8 months
* have used heroin and/or abused prescription opioids in the prior 12 months
* be 18 years of age or older at time of enrollment
* be able to provide verbal consent to participate in English

Exclusion Criteria for participants (receiving the TTIP-PRO intervention):

* demonstrate difficulty understanding the study as assessed with four true-false questions (i.e., 1. This is a research study; 2. Your participation is entirely voluntary; 3. You will be asked questions about your risk of opioid overdose.; 4. Your participation will involve several phone calls).

Inclusion Criteria for Peer Interventionists:

* be 18 years of age or older at time of enrollment
* be enrolled in a methadone-maintenance or buprenorphine- maintenance treatment program for at least one year
* report being opioid-abstinent for at least one year
* meet at least one of the following: has experienced/witnessed/lost a family member or friend to an overdose
* be able to provide informed consent in English

Exclusion criteria for Peer Interventionists:

* have significant treatment/clinical concerns as determined by treatment program staff

The primary pool of potential Peer Interventionists will be patients enrolled in the UC Health (University of Cincinnati Physicians Company) methadone-maintenance or buprenorphine- maintenance treatment programs. Recruitment will be through clinic postings and word of mouth. It is estimated that 2-3 Peer Interventionists will be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Study Acceptability (proportion of patients who: a). call about the study and b). agree to participate in the study and c). who complete the study.) | 6 months
  Acceptability of the study will be assessed based on the proportion of patients who: a). call about the study and b). agree to participate in the study and c). who complete the study.
  Acceptability of the study will be further assessed by peer interventionists who: a). complete the training and b). complete the study (i.e. continue to successfully provide intervention to assigned participants through the end of the study).

SECONDARY OUTCOMES:
Impact of TTIP-PRO on knowledge about Opioid Overdose. (will be assessed with a paired difference test (e.g., paired t-test)) | 6 months
  The impact of the TTIP-PRO on knowledge about OOD will be assessed with a paired difference test (e.g., paired t-test). Finally, summary statistics for the proportion of participants willing to be contacted by a MAT staff member after receiving the TTIP-PRO intervention will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - 3131 Harvey Avenue, Suite 104, Cincinnati, Ohio
  - UC Physicians Company, LLC Opioid Treatment Program, Cincinnati, Ohio

REFERENCES:
- [Derived] Winhusen T, Theobald J, Lewis D, Wilder CM, Lyons MS. Development and initial testing of a tailored telephone intervention delivered by peers to prevent recurring opioid-overdoses (TTIP-PRO). Health Educ Res. 2016 Apr;31(2):146-60. doi: 10.1093/her/cyw010. PMID 27004905